CLINICAL TRIAL: NCT05100823
Title: Validation of Therapeutic Efficacy Targeting the Splicing Variants in Cystic Fibrosis and CFTR Pathologies
Acronym: ONB-CFTR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrolment period completed and sufficient number of enrolments to achieve study objectives
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Foch Hospital, Suresnes, FRANCE (Unknown); Hôpital Necker-Enfants Malades (Other); Hôpital Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RECHMPL20_0423; 2020-A03529-30 (Other: ANSM)
Record Dates: First submitted 2021-09-06; First posted 2021-10-29 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Cystic Fibrosis; CFTR Gene Mutation
Keywords: genetics; cystic fibrosis; personalized therapy; Antisense OligoNucleotide strategy; splicing events; intronic variant
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nasal cells sampling and/or rectal biospy (Experimental): Depending of the patient' genotype, specific ONB-CFTR (50 nM) will be incubated at the apical face of in vitro epithelium, alone and in combination with CFTR modulators. Efficacy of ONB will be compared to a condition with oligonucleotide control incubation.
  Rectal biopsies from volunteer patients were stored as a bio-bank of organoids.
  Interventions: Procedure: Nasal cells sampling; Procedure: Rectal biopsy sampling

INTERVENTIONS:
Procedure: Nasal cells sampling — Nasal epithelium brushing in intermediate turbinate using a specific curette following a local anesthesia with Xylocaine 5% nebulizer.
Procedure: Rectal biopsy sampling — Forceps Biopsy Procedure (Servidoni et al., 2013) Only for volunteer patients included in the Montpellier center.

SUMMARY:
Cystic Fibrosis, an inherited autosomal recessive disease, arises from mutations in the CFTR gene. For intronic mutations affecting splicing events, oligonucleotides therapy has the potential to restore the production of the full length CFTR protein. Recent scientific research has demonstrated the potential of this approach to restore full length mRNA CFTR in in vitro human airway cells. The study aims to validate the therapeutic efficacy of oligonucleotide blockers (ONB) that target splicing defects associated to splicing variants in epithelia obtained from patients with Cystic Fibrosis and CFTR-related disorders.

DETAILED DESCRIPTION:
The study will include patients with various CFTR genotypes. The assessment of ONB (named ONB-CFTR) will be performed using an air-liquid interface model of airway epithelium, developed from nasal cells of patients, without or with a combination of existing CFTR modulators, depending on the patient' genotype.

This study will also aim to build a local biobank of rectal organoids from patients (only from Montpellier, France) carrying rare CFTR disease-causing variants.

ELIGIBILITY:
Inclusion Criteria:

* The subject must have given their free and informed consent and signed the consent
* The subject must be affiliated or beneficiary of a health insurance plan Women and men are included
* The patient is at least 12 years old.
* The patient has cystic fibrosis or a CFTR pathology and therefore carries two mutations (with at least one mutation affecting splicing) in the CFTR gene.
* Patients who volunteer for rectal biopsy collection (only from Montpellier University Hospital) must be at least 18 years old.

Exclusion Criteria:

* The subject is in a period of exclusion determined by a previous study.
* The subject is under judicial protection, under guardianship or under curatorship
* The subject does not accept to sign consent
* It turns out to be impossible to give informed information to the subject
* The subject does not read the French language fluently
* The subject is a pregnant or breastfeeding woman
* The subject has porphyria, or has hepatic insufficiency, or suffers from epilepsy, or suffers from conduction disorders, or suffers from severe heart failure, has a cons-indication to the use of a local anesthetic spray.

Specific non-inclusion criteria for rectal sampling:

* the subject has thrombocytopenia
* the subject has a bleeding disorder
* The patient has severe inflammation of the rectum.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-02-17 (Actual); Study Completion 2025-02-17 (Actual)

PRIMARY OUTCOMES:
Restoration of the correctly spliced CFTR mRNA (full length) using specific ONB-CFTR (designed for one splicing variant). | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  The increase will be assessed in comparison to oligonucleotide-control effect by using semi-quantitative fluorescent PCR.
Restoration of the mature CFTR protein using specific ONB-CFTR (designed for one splicing variant). | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  The increase will be assessed in comparison to oligonucleotide-control effect by using western blot
Restoration of CFTR channel function using specific ONB-CFTR (designed for one splicing variant). | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  The increase will be assessed in comparison to oligonucleotide-control effect by using electrophysiological assays (Ussing chamber).

SECONDARY OUTCOMES:
Restoration of the correctly spliced CFTR mRNA (full length) and mature CFTR protein and CFTR channel function using a pool of ONB-CFTR (a mix of specific ONB-CFTR). | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  The increase will be assessed in comparison to oligonucleotide-control effect by using semi-quantitative fluorescent PCR, western blot and electrophysiological assays (Ussing chamber).
Assessment of the amount of CFTR mRNA with normal splicing under the conditions tested. | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  That parameter will be quantified in comparison to oligonucleotide-control effect by using quantitative PCR assays.
Assessment of the amount of mature CFTR proteins under the conditions tested. | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  That parameter will be quantified in comparison to oligonucleotide-control effect by using western blot assays.
Assessment of the CFTR channel activity under the conditions tested. | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  That parameter will be quantified in comparison to oligonucleotide-control effect by using electrophysiological assays (Ussing chamber).
Increase of CFTR channel function using ONB-CFTR and CFTR modulators (correctors and/or potentiators) under the conditions tested. | 21 days after the air-liquid switch of epithelia (i.e. full differentiation)
  The increase will be assessed in comparison to oligonucleotide-control effect by using electrophysiological assays (Ussing chamber).

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France